CLINICAL TRIAL: NCT00993291
Title: Effect of Frequency Change in Bilateral Subthalamic Nucleus (STN)-DBS on Gait Function in PD
Brief Title: Deep Brain Stimulation (DBS) Frequency Effects on Gait in Parkinson's Disease(PD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Fenna Phibbs, PI, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 090873
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; DBS; Frequency; Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Baseline frequency (No Intervention): Baseline DBS frequency
  Interventions: Procedure: Frequency change to 60 Hz; Procedure: Frequency change to 130 Hz

INTERVENTIONS:
Procedure: Frequency change to 60 Hz — 60 Hz stimulation for one hour, done twice over the 5 hour study period in a randomized blinded fashion.
  Other Names: 60 Hertz
Procedure: Frequency change to 130 Hz — 130 Hz Stimulation for one hour, done twice over the 5 hour study period in a randomized blinded fashion.
  Other Names: 130 Hz

SUMMARY:
In this study the investigators will evaluate the effect of both low and high frequency Deep Brain stimulation of the subthalamic nucleus (STN) in Parkinson's patients who have noted a change in their walking. The investigators' hypothesis is:

1. Stimulation at 60 Hertz (Hz) is associated with improved gait with increased stride length and faster time on the Stand walk sit test.
2. There is no worsening of the Unified Parkinson's Disease Rating Scale (UPDRS) at 60 Hz.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient at the Vanderbilt Movement Disorders clinic.
* Report a change in their gait.
* Be able to walk independently when off PD medications for 12-16 hours.
* Have a stable dose of PD medications for the prior three months .
* Not cognitively impaired, so as to give informed consent.
* MMSE > 24.

Exclusion Criteria:

* See inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fenna T Phibbs, MD, Principal Investigator — Vanderbilt Univeristy
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Frequency: Gait analysis at the subjects baseline DBS frequency
Period: Overall Study
Arm/Group | Baseline Frequency
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Baseline Frequency
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Stride Length From Baseline
Description: Evaluation performed after DBS frequency setting changed for one hour, compared to the subject's baseline DBS frequency stride length
Time Frame: 1 hour
Measure: Mean (Full Range); unit: CM
Arm/Group | Baseline Frequency
Number analyzed (Participants) | 20
CM | 1.19 [-183 to 37]

2. Secondary Outcome: Gait Velocity
Description: gait velocity measured as change from baseline in in CM/second
Time Frame: 5 hours
Reporting Status: Not Posted

3. Secondary Outcome: Time to Walk 14 Meters
Description: Change in the time to walk 14 meters compared to baseline measured in seconds
Time Frame: 5 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Baseline Frequency
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No